CLINICAL TRIAL: NCT00830427
Title: A Phase Iib Randomised Double Blind, Placebo Controlled Parallel Group Study To Investigate The Efficacy And Safety Of Pf-00610355 Over 4 Weeks In Moderate Asthmatic Subjects.
Brief Title: A Study To Examine The Safety And Efficacy Of PF-00610355 In Moderately Asthmatic Subjects
Acronym: A7881006
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A7881006; 2008-007183-42 (EudraCT Number)
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Asthma, Bronchial; Lung Diseases, Obstructive; Respiratory Tract Diseases; Bronchial Diseases
Keywords: asthma bronchial diseases
MeSH Terms: conditions — Asthma; Lung Diseases, Obstructive; Respiratory Tract Diseases; Bronchial Diseases | interventions — N-((4'-hydroxybiphenyl-3-yl)methyl)-2-(3-(2-((-2-hydroxy-2-(4-hydroxy-3-((methylsulfonyl)amino)phenyl)ethyl)amino)-2-methylpropyl)phenyl)acetamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-00610355 (Experimental)
  Interventions: Drug: PF-00610355
- PF - 00610355 (Experimental)
  Interventions: Drug: PF - 00610355
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-00610355 — 100 mcg, QD, dry powder inhaler
  Arms: PF-00610355
Drug: PF - 00610355 — 600 mcg, QD, dry powder inhaler
  Arms: PF - 00610355
Other: Placebo — QD, dry powder inhaler
  Arms: Placebo
Drug: PF - 00610355 — 300 mcg, QD, dry powder inhaler
  Arms: PF - 00610355

SUMMARY:
This study (A7881006) is the first multiple dose study in moderate asthmatic subjects and aims to determine the safety and efficacy of PF-00610355 when subjects take PF-00610355 on a daily basis for 4 weeks in subjects maintained on inhaled corticosteroid.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a physician documented history or diagnosis of persistent asthma for at least 6 months prior to Screening Visit 1.

Trough FEV1 must be 50-100% of predicted at Screening Visit 1.

Subjects who have been maintained on a stable dose of ICS over the previous month prior to screening.

Exclusion Criteria:

* Subjects who have had a severe asthma exacerbation in the 2 months prior to screening.

Subjects meeting any of the criteria of 'very poorly controlled' according to the NIH EPR 3 guidelines.

Subjects with evidence or history of cardiovascular disease including angina, myocardial, infarction, clinically significant cardiac arrhythmia (eg, atrial fibrillation, atrial flutter,supraventricular tachycardia, ventricular tachycardia), systemic hypertension (SBP > 160 mmHg or DBP >100mmHg), pulmonary hypertension or cerebrovascular disease (including transient ischaemic attacks).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04-15 (Actual); Primary Completion 2009-12-31 (Estimated); Study Completion 2009-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline trough (24 hours post-dose) FEV1. | 4 weeks

SECONDARY OUTCOMES:
Change from baseline in heart rate. | week 0, week 4
Change from baseline in trough FEV1. | week 4
Maximum change from baseline in FEV1 from 0 to 6 hours post-dose. | week 0,week 4
Change from baseline in Asthma Quality of Life Questionnaire (AQLQ-S) score. | week 2, week 4
Pharmacokinetics of PF-00610355. | week 0, week 4

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7881006&StudyName=A%20Study%20To%20Examine%20The%20Safety%20And%20Efficacy%20Of%20PF-00610355%20In%20Moderately%20Asthmatic%20Subjects